CLINICAL TRIAL: NCT00157846
Title: Exchange of the Existing Pacemaker/ICD in Bradycardia Patients Suffering From Heart Failure to Investigate the Effect of Preventive Stimulation
Brief Title: X-Change HF - Exchange of the Existing Pacemaker/ICD in Bradycardia Patients Suffering From Heart Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to existing evidence eligible patients receive CRT treatment in first place
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CEN_G_CA_1
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure; LVEF < 35%; Bradycardia
MeSH Terms: conditions — Heart Failure; Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BiV Pacing (Experimental): Biventricular pacing for 3 months, subsequently right ventricular pacing for 3 months
  Interventions: Device: CRT-P or CRT-D Device
- RV Stimulation (Active Comparator): Right ventricular pacing for 3 months, subsequently biventricular pacing for 3 months
  Interventions: Device: CRT-P or CRT-D Device

INTERVENTIONS:
Device: CRT-P or CRT-D Device — Upgrade from ICD or pacemaker to CRT-D/CRT-P (Insync III, Insync Marquis, Insync Sentry, Insync Maximo, Concerto)

SUMMARY:
The goal of X-Change HF is to estimate the effect of biventricular stimulation in patients who need antibradycardia ventricular stimulation (more than 80%); are eligible for the exchange of an old pacemaker or implantable cardioverter defibrillator (ICD); and have ventricular dysfunction (left ventricular ejection fraction [LVEF] < 35%). All patients eligible for participation in the study will be upgraded with a cardiac resynchronization therapy (CRT)-device and receive either right ventricular or biventricular stimulation in a crossover protocol. The endpoint is functional performance measured by spiroergometry.

ELIGIBILITY:
Inclusion Criteria:

* Implanted dual-chamber pacemaker or ICD system with replacement indication

  * Because of battery end of life
  * Because of upgrade from pacemaker to ICD system

    * predominant sinus rhythm (paroxysmal atrial fibrillation [AF] < 2 hours/day)
    * predominant ventricular stimulation (>= 80%)
    * NYHA Class II-III
    * LVEF <= 35%

Exclusion Criteria:

* NYHA Class IV
* Life expectancy of less than one year because of accompanying diseases
* Myocardial infarction less than 3 months old
* Cardiac surgery less than 3 months

  * Bypass
  * Valve surgery
  * Percutaneous transluminal coronary angioplasty (PTCA)
* Thoracotomy, for implant of an epicardial LV electrode
* Medical circumstances that make participation and compliance impossible
* Patients who are not willing or able to give written consent for their study participation
* Participation in another study
* Patients less than 18 years old
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary performance measured by spiroergometry | Baseline to 7 months post-implant
  Maximal oxygen uptake (Vo2 max [ml/kg/min])

SECONDARY OUTCOMES:
Left ventricular end diastolic diameter (LVEDD [mm]) | Baseline to 7 months post-implant
N-terminal prohormone brain natriuretic peptide (NT-proBNP) [pg/ml] | Baseline to 7 months post-implant
Left ventricular ejection fraction (LVEF [%]) | Baseline to 7 months post-implant
New York Heart Association (NYHA) Class | Baseline to 7 months post-implant
Occurrence of rhythm disturbances: atrial arrhythmias (amount and duration [h/day]) | Baseline to 7 months post-implant
Occurrence of rhythm disturbances: ventricular arrhythmias (amount and duration [h/day]) | Baseline to 7 months post-implant
Heart rate variability [ms] | Baseline to 7 months post implant
Amount of hospitalizations because of heart failure (amount and duration [days]) | Baseline to 7 months post-implant
Cardiopulmonary performance measured by spiroergometry: Oxygen uptake at the anaerobic threshold (VO2 AT [s]) | Baseline to 7 months post-implant
Mortality | Baseline to 7 months post-implant

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lawo, MD, Principal Investigator — Berufsgenossenschaftliche Kliniken Bergmannsheil Bochum
Locations (10):
- Germany (10):
  - Klinikum Augsburg I. Medizinische Klinik, Augsburg
  - Charite Campus Virchow-Klinikum, Berlin
  - Unfallkrankenhaus Benjamin Franklin, Berlin
  - Ev. Freikirchliches KH Bernau und Herzzentrum Brandenburg, Bernau
  - Berufsgenossenschaftliche Kliniken Bergmannsheil, Bochum
  - Städtisches Kreiskrankenhaus, Friedrichshafen
  - Georg-August-Universität Göttingen, Göttingen
  - St.-Vincentius Klinken, Karlsruhe
  - Märkische Kliniken GmbH Klinikum Luedenscheid, Lüdenscheid
  - Krankenhaus Reinbek St. Adolf Stift, Reinbek B. Hamburg

IPD SHARING:
Plan to Share IPD: No